CLINICAL TRIAL: NCT02145494
Title: Stereotactic Prostate Augmented Radiotherapy With Cyberknife
Brief Title: The SPARC Trial: Stereotactic Prostate Ablative Radiotherapy Using Cyberknife
Acronym: SPARC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13/LO/0109; CCR 3923 (Other: Royal Marsden NHS Foundation Trust)
Record Dates: First submitted 2013-06-04; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: SBRT (stereotactic body radiotherapy); Focal boost; Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Stereotactic body radiotherapy (SBRT) to the whole prostate (36.25 Gy in 5 fractions) with a focal boost (47.5 Gy in 5 fractions) to the MRI-defined dominant tumour nodule.
  Other Names: Cyberknife

SUMMARY:
Giving a higher dose of radiation to the dominant tumour nodule within the prostate is hypothesized to improve tumour control. This trial will assess whether this technique, delivered in 5 treatments, can be delivered without increasing side effects.

DETAILED DESCRIPTION:
Aim To assess if a focal boost can be delivered to the dominant tumour nodule alongside 36.25 Gy in 5 fractions to the whole prostate gland.

Primary end-point: Acute toxicity (Radiation Therapy Oncology Group (RTOG), International prostate symptom score (IPSS))

Secondary end-points: Prostate specific antigen (PSA) nadir and 2-year biochemical control Late toxicity (IPSS, RTOG, International index of erectile function (IIEF-5)) Quality of life (EQ5D scale)

Inclusion criteria

* Prostate cancer patients with any of the following:
* PSA>20
* Gleason grade 4+3 or higher
* Stage T3a
* Exclusion criteria
* Nodal or metastatic disease
* PSA>40
* Stage T3b or higher

Study interventions

This is a phase II study which will recruit 20 patients. A dose of 36.25 Gy in 5 fractions will be delivered to the whole prostate with a simultaneous integrated boost up to 47.5 Gy in 5 fractions or to the highest dose possible within dose constraints. The boost volume will be defined on the multiparametric magnetic resonance scan by the specialist radiologist.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer patients with any of the following:

* PSA 20-40
* Gleason grade 4+3 or higher
* Stage T3a

Exclusion Criteria:

* Nodal or metastatic disease
* PSA>40
* Stage T3b or higher

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Acute genitourinary(GU) toxicity | Maximal recorded toxicity within the acute toxicity period (up to 12 weeks)
  RTOG scale acute GU toxicity will be measured at baseline, end of treatment, then 2,4 and 12 weeks post treatment. The maximal toxicity during follow up is the primary outcome measure.

SECONDARY OUTCOMES:
Acute gastrointestinal (GI) toxicity | Within 12 weeks of treatment completion
  RTOG scale
Late GI and GU toxicity | From 12 weeks until study completion
  RTOG scale
Patient reported outcomes i.e. IPSS, IIEF-5 and EQ5-D | Baseline, 12 weeks, 12 months and 6 monthly to 5 years
  IPSS, IIEF-5 and EQ5-D
Biochemical relapse-free survival | Measured at 12 weeks after completion of treatment and 3-6 monthly to 5 years thereafter
  PSA will be measured 3-6 monthly during study

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation trust, London, United Kingdom